CLINICAL TRIAL: NCT00590603
Title: Phase I/II Study of Arsenic Trioxide (Trisenox), Ascorbic Acid and Bortezomib Combination Therapy in Patients With Relapsed/Refractory Multiple Myeloma
Brief Title: Trisenox, Ascorbic Acid and Bortezomib in Patients With Relapsed/Refractory Multiple Myeloma
Acronym: AAV
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Poor accrual - terminated during Phase I; Phase II never started.
Sponsor: Duke University (Other)
Collaborators: Cephalon (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00008662; 7365 (Other: old IRB number)
Record Dates: First submitted 2007-12-26; First posted 2008-01-10 (Estimated); Last update posted 2014-01-08 (Estimated); Status verified 2012-12

CONDITIONS: Multiple Myeloma
Keywords: Multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Arsenic Trioxide; Ascorbic Acid; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Dose escalation study with two cohorts. A standard dose of Arsenic Trioxide will be given with escalating dose of Bortezomib.
  Interventions: Drug: Arsenic Trioxide, Ascorbic Acid and Bortezomib

INTERVENTIONS:
Drug: Arsenic Trioxide, Ascorbic Acid and Bortezomib — Phase I/Cohort I
  Loading:
  1. Arsenic Trioxide (ATO): 0.25 mg/kg IV over 1-2 hr qd x 5 days (Monday-Friday)
  2. Ascorbic Acid: 1000 mg by IV infusion over 15 minutes after each infusion of arsenic trioxide qd x 5 days
  Maintenance cycles (21 days)
  1. ATO: 0.25 mg/kg IV over 1-2 hr once a week x 2 weeks every 3 weeks (one cycle) for a total of 6 cycles.
  2. Ascorbic Acid 1000mg IV will be given within 30 minutes of completion of ATO.
  3. Bortezomib 1 mg/m2 is administered intravenously in a 3-5 second bolus on days 1, 8 of a 21-day cycle. ATO is given at least one hour prior to Bortezomib. The first cycle will start on week 2, after loading dose week.
  Phase I/Cohort 1 is followed by Cohort 2. Phase II uses maximum tolerated dose from Phase I.
  Other Names: AAV

SUMMARY:
This is a phase I dose escalation study to estimate the maximum tolerated dose (MTD) of the novel combination of Arsenic, Ascorbic Acid and Velcade, followed by a phase II study conducted using the MTD estimated from the phase I portion.

DETAILED DESCRIPTION:
Despite the fact the high dose therapy and autologous transplant can prolong life in patients with multiple myeloma (MM), in most studies there appears to be a continuously declining event free survival following auto-transplant indicating that few patients will be cured with this approach. A high percentage of patients the relapse in the post transplant setting will not be candidate for additional chemotherapy. We therefore, are investigating novel strategies for controlling their disease in the post transplant setting. The key theoretical issue for this study is whether concomitant Trisenox would permit the use of less toxic doses of Velcade, resulting in a less toxic but equally effective regimen.

Phase I of this study uses dose escalation to estimate the maximum tolerated dose of Arsenic, Ascorbic Acid and Velcade. Phase II is a subsequent treatment phase using the maximum tolerated dose from Phase I. In the absence of treatment delays due to adverse events, treatment may continue for 6 cycles, plus two additional cycles if patient has achieved a good response.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of relapsed/refractory multiple myeloma.
* Patients must have measurable disease, defined as localized plasmacytoma, detectable M-spike by serum protein electrophoresis (SPEP) and/or urine protein electrophoresis (UPEP), or free light chain assay, bone lytic lesions and/or bone marrow infiltration with atypical plasma-cells.
* Patients must be at least four weeks since their prior therapy. Patients will not be excluded because of any prior regimen they have received as long as they meet other requirements.
* Adequate organ function, patients with elevated creatinine due to myeloma are not excluded
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Serum potassium greater than 4.0 milliequivalent (mEq)/dL and serum magnesium greater than 1.8 mg/dL. If these electrolytes are below the specified limits on the baseline laboratory tests, supplemental electrolytes should be administered to bring the serum concentrations to these levels before administering arsenic trioxide.

Exclusion Criteria:

* Patients may not be receiving any other investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Bortezomib, Trisenox, Ascorbic acid, or other agents used in the study.
* Corrected QT interval (QTc) interval greater than 460 msec in the presence of serum potassium greater than or equal to 4.0 mEq/L and magnesium greater than or equal to 1.8 mg/dL, or underlying conduction disease that prevents measurement of the QTc interval.
* History of ventricular tachycardia or any cardiac arrhythmia requiring the placement of an automated intraventricular cardiac defibrillator or therapy with class I or class II antiarrhythmic drug.
* Ejection fraction (EF) by multigated acquisition (MUGA) scan less than 35%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Toxicity | 30 days post last dose of study drug

SECONDARY OUTCOMES:
Response | Approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Gasparetto, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States